CLINICAL TRIAL: NCT02806973
Title: A Single Center, Randomized, 4-Period Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of Single or Repeated 3 mg Doses of Intranasally Administered Glucagon in Adults With Type 1 or Type 2 Diabetes
Brief Title: A Study of Single or Repeated Doses of Glucagon in Participants With Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Locemia Solutions ULC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16428; I8R-MC-IGBG (Other: Eli Lilly and Company); AMG112 (Other: Algorithme Pharma); AGL-P5-310 (Other: Algorithme Pharma)
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nasal Glucagon (NG) - Treatment 1 (Experimental): One dose of 3 milligram (mg) NG administered in one of four study periods.
  Interventions: Drug: Nasal Glucagon
- NG - Treatment 2 (Experimental): Two NG doses, 3 mg each dose, administered 15 minutes apart, in the same nostril, in one of four study periods.
  Interventions: Drug: Nasal Glucagon
- NG - Treatment 3 (Experimental): Two NG doses, 3 mg each dose, administered 15 minutes apart, in opposite nostrils, in one of four study periods.
  Interventions: Drug: Nasal Glucagon
- NG - Treatment 4 (Experimental): Two NG doses, 3 mg each dose, administered one immediately after the other, in opposite nostrils, in one of four study periods.
  Interventions: Drug: Nasal Glucagon

INTERVENTIONS:
Drug: Nasal Glucagon — Administered intranasally.
  Other Names: AMG504-1; LY900018

SUMMARY:
This study will investigate how the body processes nasal glucagon (NG) and the effect of nasal glucagon on the body. The study is expected to last about 50 days for each participant. The study is open to adults with type 1 or type 2 diabetes and will last about 50 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with a history of Type 1 or Type 2 insulin-using diabetes of at least 1 year duration (basal only, basal bolus, meal-time only, or twice a day pre-mixed insulin)
* A female participant must meet one of the following criteria:

  * Participant is of childbearing potential and agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first administration of the study drug, during the study and for at least 30 days after the last dose of the study drug
  * Participant is of non-childbearing potential, defined as surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least 1 year without menses)
* Participant with a body mass index (BMI) greater than or equal to 18.50 kilograms per square meter (kg/m²) and below 35.00 kg/m²
* Light-, non- or ex-smokers
* In good general health with no conditions that could influence the outcome of the trial, and in the judgment of the Investigator is a good candidate for the study based on review of available medical history, physical examination and clinical laboratory evaluations

Exclusion Criteria:

* Females who are pregnant, actively attempting to get pregnant, or are lactating
* History of significant hypersensitivity to glucagon or any related products as well as severe hypersensitivity reactions (such as angioedema) to any drugs
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
* Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
* Known presence of rare hereditary problems of galactose and /or lactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Presence of clinically significant findings on nasal examination or bilateral anterior rhinoscopy, such as structural abnormalities, nasal polyps, marked septal deviation, nasal tumors
* Nasal surgery in the previous 28 days before Day 1 of this study
* Daily use of a systemic beta-blocker drug, indomethacin, warfarin or anticholinergic drugs in the previous 28 days before Day 1 of this study
* Any other concomitant maintenance therapy that would influence the outcome of the trial or compromise the safety of the participant, at the discretion of the Investigator and the Sponsor, in the previous 28 days before Day 1 of this study
* Significant history of drug dependency or alcohol abuse
* Any clinically significant illness in the previous 28 days before Day 1 of this study
* Any history of tuberculosis and/or prophylaxis for tuberculosis
* Positive urine screening of alcohol and/or drugs of abuse
* Positive results to human immunodeficiency virus (HIV) Antigen/Antibody (Ag/Ab) Combo, Hepatitis B surface Antigen (HBsAG (B) (hepatitis B)) or anti-Hepatitis C Virus (HCV (C)) tests
* Concurrent participation or intention of participating in another clinical trial during this study
* Participants who took an Investigational Product (in another clinical trial) in the previous 28 days before Day 1 of this study or who have already participated in this clinical study
* Participants who donated 50 milliliters (mL) or more of blood in the previous 28 days before Day 1 of this study
* Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before Day 1 of this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Royal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1 (T1/T2/T3/T4): Treatment 1 (T1) = Single NG dose of 3 milligram (mg), T2 = NG dose of 3 mg plus 3 mg NG dose in same nostril 15 minutes later, T3 = NG dose of 3 mg plus 3 mg NG dose in the opposite nostril 15 minutes later, T4 = NG dose of 3 mg then immediately 3 mg NG dose in the opposite nostril.
- Sequence 2 (T2/T3/T4/T1): T2 = NG dose of 3 mg plus 3 mg NG dose in same nostril 15 minutes later , T3 = NG dose of 3 mg plus 3 mg NG dose in the opposite nostril 15 minutes later, T4 = NG dose of 3 mg then immediately 3 mg NG dose in the opposite nostril, T1 = Single NG dose of 3 mg.
- Sequence 3 (T3/T4/T1/T2): T3 = NG dose of 3 mg plus 3 mg NG dose in the opposite nostril 15 minutes later, T4 = NG dose of 3 mg then immediately 3 mg NG dose in the opposite nostril, T1 = Single NG dose of 3 mg, T2 = NG dose of 3 mg plus 3 mg NG dose in same nostril 15 minutes later.
- Sequence 4 (T4/T1/T2/T3): T4 = NG dose of 3 mg then immediately 3 mg NG dose in the opposite nostril, T1 = Single NG dose of 3 mg, T2 = NG dose of 3 mg plus 3 mg NG dose in same nostril 15 minutes later, T3 = NG dose of 3 mg plus 3 mg NG dose in the opposite nostril 15 minutes later.
Period: Period 1
Arm/Group | Sequence 1 (T1/T2/T3/T4) | Sequence 2 (T2/T3/T4/T1) | Sequence 3 (T3/T4/T1/T2) | Sequence 4 (T4/T1/T2/T3)
Started | 8 | 8 | 8 | 8
Completed | 8 | 6 | 7 | 6
Not Completed | 0 | 2 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | Sequence 1 (T1/T2/T3/T4) | Sequence 2 (T2/T3/T4/T1) | Sequence 3 (T3/T4/T1/T2) | Sequence 4 (T4/T1/T2/T3)
Started | 8 | 6 | 7 | 6
Completed | 8 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 (T1/T2/T3/T4) | Sequence 2 (T2/T3/T4/T1) | Sequence 3 (T3/T4/T1/T2) | Sequence 4 (T4/T1/T2/T3)
Started | 8 | 6 | 7 | 6
Completed | 8 | 6 | 6 | 3
Not Completed | 0 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Period 4
Arm/Group | Sequence 1 (T1/T2/T3/T4) | Sequence 2 (T2/T3/T4/T1) | Sequence 3 (T3/T4/T1/T2) | Sequence 4 (T4/T1/T2/T3)
Started | 8 | 6 | 6 | 3
Completed | 8 | 6 | 6 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nasal Glucagon: All enrolled participants.
Arm/Group | Nasal Glucagon
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 32

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to T(AUC[0-tlast]) of Baseline-Adjusted Glucagon
Time Frame: -0.5, -0.25, 0.00, 0.08, 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00 hours after glucagon administration
Population: All enrolled participants with evaluable PK data.
Measure: Mean (Standard Deviation); unit: picogram*hour per millilitre (pg*hr/mL)
Groups:
- Nasal Glucagon Treatment 1: One dose of nasal glucagon.
- Nasal Glucagon - Treatment 2: Two doses of nasal glucagon, 15 minutes apart, in the same nostril.
- Nasal Glucagon - Treatment 3: Two doses of nasal glucagon, 15 minutes apart, in opposite nostrils.
- Nasal Glucagon - Treatment 4: Two doses of nasal glucagon, one immediately after the other, in opposite nostrils.
Arm/Group | Nasal Glucagon Treatment 1 | Nasal Glucagon - Treatment 2 | Nasal Glucagon - Treatment 3 | Nasal Glucagon - Treatment 4
Number analyzed (Participants) | 27 | 28 | 25 | 29
picogram*hour per millilitre (pg*hr/mL) | 2470 (1850) | 4100 (1760) | 4640 (2400) | 3610 (1880)

2. Primary Outcome: PK: Time to Maximum Concentration (Tmax) of Baseline Adjusted Glucagon
Time Frame: as for outcome 1
Population: All enrolled participants with evaluable PK data.
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | Nasal Glucagon Treatment 1 | Nasal Glucagon - Treatment 2 | Nasal Glucagon - Treatment 3 | Nasal Glucagon - Treatment 4
Number analyzed (Participants) | 27 | 28 | 25 | 29
Hour (hr) | 0.17 [0.17 to 0.75] | 0.33 [0.17 to 0.50] | 0.50 [0.17 to 0.50] | 0.33 [0.17 to 0.33]

3. Primary Outcome: PK: Maximum Change From Baseline Concentration (Cmax) of Glucagon
Time Frame: as for outcome 1
Population: All enrolled participants with evaluable PK data.
Measure: Mean (Standard Deviation); unit: picograms per millilitre (pg/mL)
Arm/Group | Nasal Glucagon Treatment 1 | Nasal Glucagon - Treatment 2 | Nasal Glucagon - Treatment 3 | Nasal Glucagon - Treatment 4
Number analyzed (Participants) | 27 | 28 | 25 | 29
picograms per millilitre (pg/mL) | 4960 (3700) | 7140 (3270) | 8080 (4170) | 6650 (3640)

4. Primary Outcome: Pharmacodynamics (PD): Area Under the Effect Concentration Time Curve (AUEC0-3) of Baseline-Adjusted Glucose From Time Zero up to 3 Hours
Time Frame: as for outcome 1
Population: All enrolled participants with evaluable PD data.
Measure: Mean (Standard Deviation); unit: Hour*millimoles per liter(hr*mmol/L)
Arm/Group | Nasal Glucagon Treatment 1 | Nasal Glucagon - Treatment 2 | Nasal Glucagon - Treatment 3 | Nasal Glucagon - Treatment 4
Number analyzed (Participants) | 27 | 28 | 25 | 29
Hour*millimoles per liter(hr*mmol/L) | 157 (95.7) | 168 (99.3) | 190 (95.3) | 194 (117)

5. Primary Outcome: PD: Time to Maximum Concentration (Tmax) of Baseline-Adjusted Glucose
Time Frame: as for outcome 1
Population: All enrolled participants with evaluable PD data.
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | Nasal Glucagon Treatment 1 | Nasal Glucagon - Treatment 2 | Nasal Glucagon - Treatment 3 | Nasal Glucagon - Treatment 4
Number analyzed (Participants) | 27 | 28 | 25 | 29
Hour (hr) | 0.75 [0.50 to 1.50] | 1.00 [0.50 to 2.50] | 1.00 [0.75 to 1.75] | 1.00 [0.50 to 2.50]

6. Primary Outcome: PD: Baseline-Adjusted Glucose Maximum Concentration (BGmax)
Time Frame: as for outcome 1
Population: All enrolled participants with evaluable PD data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nasal Glucagon Treatment 1 | Nasal Glucagon - Treatment 2 | Nasal Glucagon - Treatment 3 | Nasal Glucagon - Treatment 4
Number analyzed (Participants) | 27 | 28 | 25 | 29
mmol/L | 89.5 (36.6) | 98.4 (39.4) | 108 (36.9) | 105 (44)

7. Other Pre Specified Outcome: PK: Area Under the Curve Extrapolated to Infinity (AUC[0-inf]) of Glucagon
Time Frame: as for outcome 1
Population: All enrolled participants with evaluable PK data.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Nasal Glucagon Treatment 1 | Nasal Glucagon - Treatment 2 | Nasal Glucagon - Treatment 3 | Nasal Glucagon - Treatment 4
Number analyzed (Participants) | 27 | 28 | 25 | 29
pg*hr/mL | 2730 (1860) | 4440 (1800) | 4940 (2400) | 3900 (1920)

ADVERSE EVENTS:
Time Frame: First dose of study drug (Day 1) until post-study completion (Day 50)
Arm/Group | Nasal Glucagon Treatment 1 | Nasal Glucagon - Treatment 2 | Nasal Glucagon - Treatment 3 | Nasal Glucagon - Treatment 4
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28 | 0/25 | 1/29
Other Adverse Events (participants affected / at risk) | 27/27 | 28/28 | 25/25 | 27/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Glucagon Treatment 1 (N=27) | Nasal Glucagon - Treatment 2 (N=28) | Nasal Glucagon - Treatment 3 (N=25) | Nasal Glucagon - Treatment 4 (N=29)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Glucagon Treatment 1 (N=27) | Nasal Glucagon - Treatment 2 (N=28) | Nasal Glucagon - Treatment 3 (N=25) | Nasal Glucagon - Treatment 4 (N=29)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 2 (2) | 5 (5) | 2 (2) | 3 (3)
Eye pain (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Lacrimation increased (Eye disorders) | 25 (25) | 25 (38) | 23 (36) | 25 (27)
Ocular hyperaemia (Eye disorders) | 2 (2) | 5 (6) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 9 (10) | 5 (5) | 9 (9)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 7 (7) | 3 (3) | 3 (3)
Asthenia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vessel puncture site bruise (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 3 (3) | 4 (6) | 3 (3) | 4 (7)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulse abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 6 (7) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 9 (10) | 14 (15) | 12 (14) | 12 (12)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2)
Parosmia (Nervous system disorders) | 2 (2) | 2 (2) | 3 (4) | 4 (4)
Sinus headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) | 2 (2) | 2 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (3) | 2 (2) | 3 (3)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (12) | 6 (8) | 10 (12)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6) | 5 (7) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (4) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days